CLINICAL TRIAL: NCT03474926
Title: Prospective Randomized Phase II Trial: Comparing the Prognostic Value of Routine Lymphadenectomy Versus Lymphadenectomy Only for Lymph Nodes Enlargement Found in Preoperative Imaging or During Surgery Undergoing Nephroureterectomy in Patients With Primary Upper Tract Urothelial Carcinoma
Brief Title: Prognostic Value of Lymph Node Dissection in Patients With Transitional Cell Carcinoma of the Upper Urinary Tract
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTUC-LND collaboration 1
Record Dates: First submitted 2018-02-27; First posted 2018-03-23 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Lymph Node Dissection
Keywords: urothelial cancer; nephroureterectomy; Upper urinary tract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine lymph node dissection (LND) during nephroureterectomy (Experimental): Template-based LND was carried out in all patients in this group. The anatomical extent of LND is described in previous study. Lymph node specimens were sampled "en bloc" with surrounding adipose tissue, and were sent to pathological examination as individual packets with the surrounding adipose tissue.
  Interventions: Procedure: Routine Template-based lymphadenectomy
- LND for lymph nodes enlargement found before or during surgery (Active Comparator): LND was carried out only in patients who have lymph nodes enlargement in preoperative imaging (CTU or enhanced MRI) or who were found lymph nodes enlargement during surgery.
  Interventions: Procedure: LND only for lymph nodes enlargement found in preoperative image or during surgery

INTERVENTIONS:
Procedure: Routine Template-based lymphadenectomy — Template-based LND was carried out in all patients in this group. The anatomical extent of LND is described in previous study. Lymph node specimens were sampled "en bloc" with surrounding adipose tissue, and were sent to pathological examination as individual packets with the surrounding adipose tissue.
  Arms: Routine lymph node dissection (LND) during nephroureterectomy
Procedure: LND only for lymph nodes enlargement found in preoperative image or during surgery — LND was carried out only in patients who have lymph nodes enlargement in preoperative imaging (e.g. CTU or enhanced MRI) or who were found lymph nodes enlargement during surgery
  Arms: LND for lymph nodes enlargement found before or during surgery

SUMMARY:
Recent studies showed the therapeutic benefit of lymphadenectomy in advanced stage urothelial carcinoma of the upper urinary tract, but there is still a lack of prospective studies. Thus, the current guideline recommends lymph node dissection for invasive upper tract urothelial carcinoma (UTUC) on the basis of insufficient evidence. Also, the preoperative judgment of muscle invasive pathological stage T 2+,or N+ is difficult from preoperative imaging. In the investigators' clinical practice, the surgeons performed dissection of regional lymph nodes only in patients with enlargement of lymph nodes found in preoperative imaging or during surgery. The aim of this multi-institutional study was to examine the role of lymphadenectomy in urothelial carcinoma of the upper urinary tract.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with upper tract urothelial carcinoma
* have no distant metastasis
* have an Eastern Cooperative Oncology Group (ECOG) score 0 to 2
* expected to receive radical nephroureterectomy

Exclusion Criteria:

* a prior history of bladder cancer
* administration of neoadjuvant chemotherapy
* deny to receive long term follow-up
* patients with contralateral UTUCs
* patients with synchronous muscle invasive bladder cancer

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 36 month
  Disease free survival rate in the 36 month following nephroureterectomy

SECONDARY OUTCOMES:
Cancer specific survival | 36 month
  Cancer specific survival rate in the 36 month following nephroureterectomy
Overall survival | 36 month
  Overall survival rate in the 36 month following nephroureterectomy
The recurrence rate of bladder cancer in the 36 month following nephroureterectomy | 36 month
  The recurrence rate of bladder cancer in the 36 month following nephroureterectomy
Perioperative complications rate | 90 day
  Perioperative complications were evaluated up to 90 days after surgery, and were graded by Clavien-Dindo classiﬁcation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xue, M.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Liqun Zhou, M.D, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijin, Beijin
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality